CLINICAL TRIAL: NCT04564248
Title: Setting up a Website in Paediatric Surgery at the Rouen University Hospital for Parents and Children to Better Understand the Postoperative Prescription of Painkillers.
Acronym: DOLIPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/0045/HP
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Paediatric Surgery; Analgesics Prescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- website access for families (Experimental)
  Interventions: Other: Website access
- standard care (No Intervention)

INTERVENTIONS:
Other: Website access — website access will be provide to families
  Arms: website access for families

SUMMARY:
Although outpatient surgery is increasing in France, particularly in paediatrics, compliance with analgesics prescriptions and pain management on return home remain poorly controlled parameters, although they are essential for optimal care. This is due, among other things, to parents' lack of knowledge and fears about the medicines prescribed to them. The paediatric anaesthesia unit of the Rouen University Hospital has set up a website for families to improve understanding of and compliance with the prescription of painkillers and thus improve the management of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a Physical status score equal or II
* Ages 2-12
* Receiving outpatient surgery according to the eligibility criteria established in the latest expert recommendations in 2009 and in accordance with the service's practices

Exclusion Criteria:

* Lack of access to internet
* Cognitive dysfunction in children that interfere with understanding instructions
* Patient already receiving a analgesic treatment

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Number of analgesic treatment taken | day 1 after surgery

SECONDARY OUTCOMES:
Number of analgesic treatment taken | day 2 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DELMON, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France